CLINICAL TRIAL: NCT04752527
Title: The Clinical Study of Individualized Induction Therapy for Non-elderly Patients With Acute Myeloid Leukemia and Adverse Risk Features Guided by Rapid Screening With FISH and NGS
Brief Title: Individualized Induction Therapy for Non-elderly Acute Myeloid Leukemia Patients With Adverse Risk Features
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-AML01
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment regime (Experimental): combination of venetoclax plus azacitidine, and Sorafenib for patients with high FLT3-ITD allelic ratio
  Interventions: Drug: venetoclax combined with decitabine

INTERVENTIONS:
Drug: venetoclax combined with decitabine — combination of venetoclax plus decitabine, and sorafenib for patients with high FLT3-ITD allelic ratio. (On day 1 of cycle 1, decitabine 20 mg/m2 will be given intravenously, and will continue for 5 days. Simultaneously the patient will start out with Venetoclax 100mg and progress to 400mg until the 28 day cycle is finished. For patients with high FLT3-ITD allelic ratio, sorafenib was administered at a dose of 400mg orally twice daily, on days 3 through 28.
  Other Names: combination of venetoclax plus decitabine with or without sorafenib

SUMMARY:
Individualized induction therapy will be applied to the non-elderly acute myeloid leukemia (AML) patients with adverse genetic risk features guided by rapid screening with fluorescence in situ hybridization (FISH) and next-generation sequencing (NGS), such as the combination of Venetoclax plus decitabine, and Sorafenib for patients with high (FMS)-like tyrosine kinase 3-internal tandem duplication (FLT3-ITD) allelic ratio. This study aims to improve induction therapy for non-elderly AML patients with adverse genetic risk features, reduce treatment-related complications, and improve overall survival.

DETAILED DESCRIPTION:
The non-elderly AML patients who meet the adverse risk group defined as 2017 European LeukemiaNet (ELN) risk stratification, are more likely to be refractory to intensive induction and have low rates of long-term survival. Venetoclax (drug name) plus decitabine or azacitidine showed tolerable safety and favorable overall response rate (ORR )(complete remission (CR)+CR with incomplete hematologic recovery (CRi) rate: 67%) in elderly AML patients. In addition, combination therapy with sorafenib, cytarabine and idarubicin was able to induce a high CR rate in non-elderly AML patients with FLT3 mutations and a 1-year probability of survival of 74%. The fast next-generation sequencing together with FISH can identify the adverse genetic risk features in AML patients within 72 hours. Individualized induction therapy will be applied to the non-elderly AML patients with adverse genetic risk features guided by rapid screening with FISH and NGS, such as the combination of venetoclax plus decitabine, and Sorafenib for patients with high FLT3-ITD allelic ratio. This study aims to improve induction therapy for non-elderly AML patients with adverse genetic risk features, reduce treatment-related complications, and improve overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 59 > =Age (years) >= 18;
2. Newly diagnosed as AML patients according to World Health Organization (WHO) classification;
3. AML patients meet the adverse risk group according to 2017 European Leukemia Net risk stratification;
4. Patients have not received prior therapy for AML (except HU);
5. Eastern Cooperative Oncology Group (ECOG) Performance status of 0,1, 2 ;
6. Liver function: Total bilirubin ≦3 upper limit of normal (ULN); aspartate aminotransferase (AST) ≦3 ULN; alanine aminotransferase (ALT)≦3 ULN(except extramedullary infiltration of leukemia)
7. Renal function：Ccr ≧30 ml/min;
8. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Acute promyeloid leukemia；
2. AML with central nervous system (CNS) infiltration；
3. Patients have received prior hypomethylating agents (HMA) therapy for myelodysplastic syndrome (MDS) and progressed to AML；
4. HIV infection;
5. Patients with severe heart failure (grade 3-4) ;
6. Evidence of other clinically significant uncontrolled condition(s) including, but not limited to: a) Uncontrolled and/or active systemic infection (viral, bacterial or fungal); b) Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. c)An active second cancer that requires treatment within 6 months of study entry
7. Patients deemed unsuitable for enrolment by the investigator;
8. Patients willing to receive intensive induction chemotherapy
9. Female who are pregnant, breast feeding or childbearing potential without a negative urine pregnancy test at screen；
10. Patients reject to participate in the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
CR/CRi/morphologic leukemia free state (MLFS) | Study start date to study end date, or death, whichever comes first, up to 4 years
  Complete remission/complete remission with incomplete count recovery/Morphologic Leukemia Free State（after one cycle or two cycles of induction therapy）

SECONDARY OUTCOMES:
Event Free Survival(EFS) | Study start date to study end date, or death, whichever comes first, up to 4 years
  Event Free Survival
Overall Survival(OS) | Study start date to study end date, or death, whichever comes first, up to 4 years
  Overall Survival
Incidence of Adverse Events | Study start date to study end date, or death, whichever comes first, up to 4 years
  infection, blood transfusion, and other toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Jiangsu Institute of Hematology, Suzhou, Jiangsu, China